CLINICAL TRIAL: NCT01513356
Title: Evaluation of PI3K/AKT/mTOR Signaling Pathway Using BKM120 in Early Breast Cancer
Brief Title: Pharmacodynamic Study of BKM120 in Breast Cancer
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Sofia Perea, Director Clinical Trials Unit. (Other)
Collaborators: Novartis (Industry)
Responsible Party: Sponsor-Investigator, Sofia Perea, Director Clinical Trials Unit., Director Clinical Research Unit, Grupo Hospital de Madrid
Organization: Grupo Hospital de Madrid (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: CBKM120XES01T
Record Dates: First submitted 2011-12-21; First posted 2012-01-20 (Estimated); Last update posted 2014-04-02 (Estimated); Status verified 2014-04

CONDITIONS: Breast Cancer
Keywords: breast; cancer; BKM120
MeSH Terms: conditions — Breast Neoplasms; Neoplasms | interventions — NVP-BKM120

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- CBKM120 (Experimental): BKM120 will be administered on a continuous once daily dosing schedule at a dose of 100 mg (p.o.)during 28 days
  Interventions: Drug: BKM120

INTERVENTIONS:
Drug: BKM120 — BKM120 will be administered on a continuous once daily dosing schedule at a dose of 100 mg (p.o.)until progression of disease or unacceptable toxicity or a maximum of 4 weeks.

SUMMARY:
BKM120 is a potent and highly specific oral pan-class I phosphatidylinositol-3-kinase (PI3K) inhibitor, currently under investigation in a first-in-man study in patients with advanced solid tumors (wild type and PIK3CA-mutated). Consistent, dose-dependent pharmacodynamic activity has been demonstrated and clear signs of anti-tumor activity have been seen with BKM120.

DETAILED DESCRIPTION:
BKM120 is a potent and highly specific oral pan-class I phosphatidylinositol-3-kinase (PI3K) inhibitor, currently under investigation in a first-in-man study in patients with advanced solid tumors (wild type and PIK3CA-mutated). Consistent, dose-dependent pharmacodynamic activity has been demonstrated and clear signs of anti-tumor activity have been seen with BKM120. Three breast cancer patients showed significant tumor shrinkage after ≥ 2 months. Two confirmed partial responses (PRs) per RECIST have been seen, one in a patient with a triple negative KRAS-mutated breast cancer and the other in a patient with an estrogen receptor (ER)-positive, PIK3CAmutated tumor. Two minor responses have also been observed; one of these occurred in a HER2+/ER+ breast cancer patient.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* ER+ / HER2 negative breast cancer patients
* WHO performance status £ 2
* Previously untreated histologically confirmed invasive, non-metastatic, breast carcinoma with a tumor size ≥ 1,5cm and non urgent surgical treatment
* Activated Pi3K pathway in breast cancer trucut biopsy
* Documentation of negative pregnancy test for patients of child bearing potential within 7 days prior to start study treatment. Sexually active pre-menopausal patients must use adequate contraceptive measures, excluding estrogen containing contraceptives, while on study.
* Patients must meet the following laboratory criteria within 7 days prior to start the study treatment:
* Hematology
* Neutrophil count of > 1200/mm3
* Platelet count of > 100,000/ mm3
* Hemoglobin > 90g/L
* Biochemistry
* AST/SGOT and ALT/SGPT < 2.5 x upper limit of normal (ULN) or < 5.0 x ULN if the transaminase elevation is due to liver metastases
* Total bilirubin < 1.5 x ULN [Patients with Gilbert Syndrome must have total bilirubin < 3 ULN]
* Cholesterol < ULN - 7.75 mmol/L and Triglycerides < ULN - 2.5 x ULN (with lipid-lowering drugs permitted)
* Serum creatinine < 1.5 x ULN or 24-hour creatinine clearance > 60 mL/min
* Serum albumin > LLN or > 30 g/L
* Fasting plasma glucose ≤ 140 mg/dL (7.8 mmol/L)

Exclusion Criteria:

* Patients who have received prior treatment with a P13K inhibitor
* Patients with a known hypersensitivity to BKM120 or to its excipients
* Patients with a history of photosensitivity reactions to other drugs
* Patients with the following mood disorders as judged by the Investigator or a psychiatrist, or as result of patient's mood assessment questionnaire:
* Medically documented history of or active major depressive episode, bipolar disorder (I or II), obsessive-compulsive disorder, schizophrenia, a history of suicidal attempt or ideation, or homicidal ideation (immediate risk of doing harm to others)
* ≥ CTCAE grade 3 anxiety The psychiatric judgment overrules the mood assessment questionnaire result/investigators judgment.
* Impairment of gastrointestinal (GI) function or GI disease that may significantly alter the absorption of BKM120 (e.g., ulcerative diseases, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome, or small bowel resection). Patients with unresolved diarrhea will be excluded as previously indicated
* Patients with diabetes mellitus requiring insulin treatment, history of gestational diabetes mellitus
* Impaired cardiac function or clinically significant cardiac diseases
* LVEF < 45% as determined by MUGA scan or ECHO
* Complete left bundle branch block
* ST depression or elevation of ≥ 1.5 mm in 2 or more leads
* Congenital long QT syndrome
* History or presence of ventricular arrhythmias or atrial fibrillation
* Clinically significant resting bradycardia (< 50 beats per minute)
* QTc > 460 msec on screening ECG
* Right bundle branch block + left anterior hemiblock (bifascicular block)
* Unstable angina pectoris ≤ 3 months prior to starting the study drug
* Acute myocardial infarction ≤ 3 months prior to starting the study drug
* Other clinically significant heart disease such as congestive heart failure requiring treatment or uncontrolled hypertension
* Patients who have been treated with any hematopoietic colony-stimulating growth factors (e.g., G-CSF, GM-CSF) ≤ 2 weeks prior to starting study drug. Erythropoietin or darbepoetin therapy, if initiated before enrollment, may be continued
* Patients who are currently receiving treatment with medication that has the potential to prolong the QT interval or inducing Torsades de Pointes and the treatment cannot either be discontinued or switched to a different medication prior to starting study drug
* Patients who are currently receiving treatment with therapeutic doses of warfarin sodium (Coumadin®)
* Patients with known coagulopathies
* Patients who have received chemotherapy, immunotherapy (except for trastuzumab) or investigational drugs ≤ 4 weeks prior to starting study drug or who have not recovered from side effects of such therapy
* Patients who have received any continuous-dosing (i.e. daily dosing, ever-other-day dosing, Monday-Wednesday-Friday dosing weekly etc) therapeutic modalities or investigational drug (excluding monoclonal antibodies) ≤ 5 half lives prior to starting study drug or who have not recovered from side effects of such therapy
* Patients who have received corticosteroids ≤ 2 weeks prior to starting study drug or who have not recovered from the side effects of corticosteroid treatment
* Patients who have received wide field radiotherapy ≤ 4 weeks or limited field radiation for palliation ≤ 2 weeks prior to starting study drug or who have not recovered from side effects of such therapy.
* Patients who have undergone major surgery ≤ 2 weeks prior to starting study drug or who have not recovered from side effects of such therapy
* Women of child-bearing potential who are pregnant or breast feeding and adults of reproductive potential not employing an effective method of birth control. Adequate contraception must be used throughout the trial and for 8 weeks after the last dose of study drug, by both sexes. Women of child-bearing potential must have a negative serum pregnancy test ≤ 7 days prior to starting BKM120
* Male patients whose sexual partner(s) are WOCBP who are not willing to use adequate contraception, during the study and for 8 weeks after the end of treatment
* Patients with a known diagnosis of human immunodeficiency virus (HIV) infection (HIV testing is not mandatory)
* Patients with a history of another primary malignancy that is currently clinically significant, has potential for metastases or currently requires active intervention
* Patients who have any severe and/or uncontrolled medical conditions or other conditions that could affect their participation in the study such as:
* Patients with any other concurrent severe and/or uncontrolled concomitant medical conditions (e.g. active or uncontrolled infection) that could cause unacceptable safety risks or compromise compliance with the protocol
* History of noncompliance to medical regimens
* Patients unwilling to or unable to comply with the protocol

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2012-10; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
- To determine the grade of inhibition of PI3K/mTOR pathways, in pre-surgery setting with BKM120 | 28 days
  Biomarkers assessments must be performed at baseline and at the end of study treatment. The following biomarkers will be assessed: PI3K, KRAS, pAkt and -RPS6p

SECONDARY OUTCOMES:
Number, grade and relationship of adverse events with BKM120 | 28 days
Potential predictive biomarkers (PI3K mutation, KRAS, pAkt and RPS6p) for a pathologic complete response relating to BKM120 | 28 days

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Madrid Norte Sanchinarro- CIOCC, Madrid, Madrid, Spain

REFERENCES:
- [Background] Bendell JC, Rodon J, Burris HA, de Jonge M, Verweij J, Birle D, Demanse D, De Buck SS, Ru QC, Peters M, Goldbrunner M, Baselga J. Phase I, dose-escalation study of BKM120, an oral pan-Class I PI3K inhibitor, in patients with advanced solid tumors. J Clin Oncol. 2012 Jan 20;30(3):282-90. doi: 10.1200/JCO.2011.36.1360. Epub 2011 Dec 12. PMID 22162589
- [Background] Park E, Park J, Han SW, Im SA, Kim TY, Oh DY, Bang YJ. NVP-BKM120, a novel PI3K inhibitor, shows synergism with a STAT3 inhibitor in human gastric cancer cells harboring KRAS mutations. Int J Oncol. 2012 Apr;40(4):1259-66. doi: 10.3892/ijo.2011.1290. Epub 2011 Dec 8. PMID 22159814
- [Background] Koul D, Fu J, Shen R, LaFortune TA, Wang S, Tiao N, Kim YW, Liu JL, Ramnarian D, Yuan Y, Garcia-Echevrria C, Maira SM, Yung WK. Antitumor activity of NVP-BKM120--a selective pan class I PI3 kinase inhibitor showed differential forms of cell death based on p53 status of glioma cells. Clin Cancer Res. 2012 Jan 1;18(1):184-95. doi: 10.1158/1078-0432.CCR-11-1558. Epub 2011 Nov 7. PMID 22065080
- [Background] Maira SM. PI3K inhibitors for cancer treatment: five years of preclinical and clinical research after BEZ235. Mol Cancer Ther. 2011 Nov;10(11):2016. doi: 10.1158/1535-7163.MCT-11-0792. No abstract available. PMID 22072802
- [Background] Leung E, Kim JE, Rewcastle GW, Finlay GJ, Baguley BC. Comparison of the effects of the PI3K/mTOR inhibitors NVP-BEZ235 and GSK2126458 on tamoxifen-resistant breast cancer cells. Cancer Biol Ther. 2011 Jun 1;11(11):938-46. doi: 10.4161/cbt.11.11.15527. Epub 2011 Jun 1. PMID 21464613
- [Background] Brunner-Kubath C, Shabbir W, Saferding V, Wagner R, Singer CF, Valent P, Berger W, Marian B, Zielinski CC, Grusch M, Grunt TW. The PI3 kinase/mTOR blocker NVP-BEZ235 overrides resistance against irreversible ErbB inhibitors in breast cancer cells. Breast Cancer Res Treat. 2011 Sep;129(2):387-400. doi: 10.1007/s10549-010-1232-1. Epub 2010 Nov 3. PMID 21046231
- [Background] Brachmann SM, Hofmann I, Schnell C, Fritsch C, Wee S, Lane H, Wang S, Garcia-Echeverria C, Maira SM. Specific apoptosis induction by the dual PI3K/mTor inhibitor NVP-BEZ235 in HER2 amplified and PIK3CA mutant breast cancer cells. Proc Natl Acad Sci U S A. 2009 Dec 29;106(52):22299-304. doi: 10.1073/pnas.0905152106. Epub 2009 Dec 10. PMID 20007781
- [Background] Maira SM, Stauffer F, Brueggen J, Furet P, Schnell C, Fritsch C, Brachmann S, Chene P, De Pover A, Schoemaker K, Fabbro D, Gabriel D, Simonen M, Murphy L, Finan P, Sellers W, Garcia-Echeverria C. Identification and characterization of NVP-BEZ235, a new orally available dual phosphatidylinositol 3-kinase/mammalian target of rapamycin inhibitor with potent in vivo antitumor activity. Mol Cancer Ther. 2008 Jul;7(7):1851-63. doi: 10.1158/1535-7163.MCT-08-0017. Epub 2008 Jul 7. PMID 18606717